CLINICAL TRIAL: NCT06153823
Title: Effectiveness of Virtual Reality Glasses Integrated With Sign Language on Dental Anxiety Among Children With Hearing Impairment During Pulpotomy Procedure (Randomized Controlled Clinical Trial)
Brief Title: Virtual Reality Glasses Integrated With Sign Language on Dental Anxiety Among Children With Hearing Impairment During Pulpotomy Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0665-04/2023
Record Dates: First submitted 2023-11-11; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Dental Anxiety

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality glasses (Experimental)
  Interventions: Other: virtual reality glasses
- show-tell-do technique. (Active Comparator)
  Interventions: Other: Tell Show and Do

INTERVENTIONS:
Other: virtual reality glasses — child behavior management will be done by using VR glasses distraction
  Arms: virtual reality glasses
Other: Tell Show and Do — child behavior management will be done by using tell show and do technique
  Arms: show-tell-do technique.

SUMMARY:
To evaluate the impact of using virtual reality glasses using sign language as a distraction method to reduce the dental anxiety in moderate to severe hearing-impaired children compared to the conventional behavior management technique during pulpotomy treatment.

The study will be a randomized controlled parallel two arms clinical trial, a total of 40 healthy children aged 5-7 years with moderate to severe hearing disability, will be selected from Pediatric Dentistry and dental public health Department, Faculty of Dentistry, Alexandria University, Egypt. Children selected should have at least one primary molar indicated for pulpotomy. The eligible participants will be randomly assigned to one of two groups: the study group, which will use virtual reality glasses with sign language as a distraction method to manage children's behavior, and the control group, which will use the conventional behavior management strategies including show-tell-do, and positive reinforcement. Local anesthesia will be given and pulpotomy procedure will be done on the selected tooth followed by stainless steel crown restoration. Pre and post-operative assessment of child's dental anxiety will be done using three methods: physiologically using pulse oximeter for measuring the heart rate, objectively using Venham clinical anxiety rating scale, and subjectively using the modified facial image scale.

ELIGIBILITY:
Inclusion Criteria:

* Children with Frankl behavior rating score 2 or 3.
* Children requiring pulpotomy in one of their primary molars.
* Parents who accepted to give their consent and participate in the study.

Exclusion Criteria:

* Children with any medical condition other than hearing disability (ASA II, III & IV).
* Syndromic children with hearing impairment.
* Children with previous bad dental experience.

Ages: 5 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in child anxiety level | up to 2 months
  This objective measure scores the child's level of anxiety with a correlating behavior description It consists of 6 categories (range from 0 to 5) where 0= relaxed, 1=uneasy, 2= tense, 3= reluctant, 4= interference, 5= out of contact.

SECONDARY OUTCOMES:
Change in heart rate | up to 2 months
  Heart rate (HR) is a physiological sign of pain. It will be measured using a pulse oximeter
Change in child anxiety level by subjective method | up to 2 months
  A modified face scale will be used to subjectively record anxiety . It consists of three schematic faces with different facial expressions for happy and sad faces representing: (A) satisfaction; (B) indifference; and (C) dissatisfaction, respectively

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt

REFERENCES:
- [Derived] Salama RM, El-Habashy LM, Zeitoun SI. Effectiveness of virtual reality glasses with integrated sign language in reducing dental anxiety during pulpotomy in children with hearing impairment: a randomized controlled trial. BMC Oral Health. 2024 Nov 15;24(1):1388. doi: 10.1186/s12903-024-05129-1. PMID 39548423